CLINICAL TRIAL: NCT05758298
Title: Assessing the Use of Nicotine Gum to Decrease Betel Nut Chewing in Saipan
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Have not received IRB approval.
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Commonwealth Healthcare Corporation (Other)
Responsible Party: Principal Investigator, Mary Chang, ASSOC PROFESSOR, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: STU-2022-1040
Record Dates: First submitted 2023-02-24; First posted 2023-03-07 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Betel Nut Cessation
Keywords: replacement therapy
MeSH Terms: interventions — Nicotine; Chewing Gum

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Consenting research team members will not know the order of the randomization schedule or what numbers correspond to treatment options. Blinded members of the research team will receive the participants chew logs for analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Non-medicated gum Arm (Placebo Comparator): Participants in this group will receive the non-medicated gum in mint flavor.
  Interventions: Other: Non-medicated gum
- Nicotine 2mg gum Arm (Experimental): Participants in this group will receive the 2mg Nicotine gum in mint flavor.
  Interventions: Drug: NICOTINE 2MG GUM
- Nicotine 4mg gum Arm (Experimental): Participants in this group will receive the 4mg Nicotine gum in mint flavor.
  Interventions: Drug: NICOTINE 4MG GUM

INTERVENTIONS:
Other: Non-medicated gum — Non-medicated, regular chewing gum in mint flavor (6 pieces of gum per day given, but used as needed).
  Arms: Non-medicated gum Arm
Drug: NICOTINE 2MG GUM — Nicotine 2mg chewing gum in mint flavor (6 pieces of gum per day given, but used as needed).
  Arms: Nicotine 2mg gum Arm
Drug: NICOTINE 4MG GUM — Nicotine 4mg chewing gum in mint flavor (6 pieces of gum per day given, but used as needed).
  Arms: Nicotine 4mg gum Arm

SUMMARY:
The study will include a prospective, randomized, double-blinded trial, with a total of 45 subjects enrolled. Research subjects will be recruited from a population of adult patients (current patients at Commonwealth Healthcare Corporation) 18 years or older who are daily betel nut chewers who add tobacco to their chew. One of the study team members will be traveling to Commonwealth of Northern Mariana Islands and a letter of support has been obtained in order to conduct the study.

Eligible patients must be non-tobacco smokers, be actively interested in betel nut reduction or cessation, and chew at least four times a day on average. Subjects will be randomized equally into three distinct groups for the purpose of this study:

* non-medicated regular chewing gum
* nicotine 2 mg gum
* nicotine 4 mg gum

DETAILED DESCRIPTION:
Objectives include:

A. Assess the efficacy of nicotine gum as a replacement therapy in reducing betel nut usage among adult betel nut chewers in Saipan.

B. Determine if larger doses of nicotine in gum are associated with statistically significantly greater reductions in betel nut usage.

C. Leverage results from this study as a means to explore further if nicotine gum would be helpful in decreasing betel nut consumption.

ELIGIBILITY:
Inclusion Criteria:

* Daily betel nut chewers who use betel nut and tobacco in their chews.
* Interested in betel nut reduction or cessation when they are informed of the study.
* Must chew greater than or equal to 4 times a day.
* Must have an appointment with a provider at the Commonwealth Healthcare Corporation

Exclusion Criteria:

* Tobacco smokers
* Under the age of 18 years old
* Potential subjects unable to accurately estimate the number of average betel nut chews per day (will be able to re-present for enrollment if they are able to make an accurate estimate of chews per day after keeping a personal record chew for one week or more)
* Pregnant patients
* Established diagnosis of oropharyngeal cancer

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in average "betel nut chews per day" at 3 months | Baseline, 3 months
  Average "betel nut chews per day" will be calculated by taking average of one full week of self-reported daily chews

CONTACTS AND LOCATIONS:
Overall Officials: Mary Chang, MD, Principal Investigator — University of Texas Southwestern Medical Center

IPD SHARING:
Plan to Share IPD: No